CLINICAL TRIAL: NCT04193085
Title: Wearable Technology to Assess Gait Function in Spinal Muscle Atrophy and Duchenne Muscular Dystrophy
Brief Title: Wearable Technology to Assess Gait Function in SMA and DMD
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Muscular Dystrophy Association (Other); Stevens Institute of Technology (Other)
Responsible Party: Principal Investigator, Jacqueline Montes, Assistant Professor of Rehabilitation and Regenerative Medicine , Rehab & Regenerative Med PT, Columbia University
Other Study IDs: AAAS5641
Record Dates: First submitted 2019-11-11; First posted 2019-12-10 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-02

CONDITIONS: Spinal Muscular Atrophy Type 3; Duchenne Muscular Dystrophy
Keywords: Spinal Muscular Atrophy; SMA; Duchenne Muscular Dystrophy; DMD; instrumented insole; neuromuscular disease; six minute walk test; machine learning model; gait analysis; wearable; ambulatory; stride; foot-worn
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal; Neuromuscular Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Spinal Muscular Atrophy (SMA): ambulatory children and adults at least 5 years old by the time of enrollment with genetically confirmed SMA
  Interventions: Other: Observational
- Duchenne / Becker Muscular Dystrophy (DMD/BMD): ambulatory children and adults ages at least 5 years old by the time of enrollment with genetically confirmed Duchenne or Becker muscular dystrophy or evidence on muscle biopsy with a clinical presentation consistent with DMD /BMD.
  Interventions: Other: Observational
- Healthy Control: The healthy control group will be age and gender-matched to the SMA and DMD groups as best as possible
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The purpose of this project is to devise instrumented insoles capable of accurately measuring gait at each footfall, over multiple hours in any environment. To achieve high accuracy, the investigators will develop a new learning-based calibration framework. Features will be tested in controlled lab settings 39 during a single visit in people with SMA (13), DMD (13) and healthy controls (13) and in 15 participants in real-life environments.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) and Duchenne muscular dystrophy (DMD) are genetic disorders that often result in progressive weakness and impaired function. Results from this study will help characterize how gait is affected in SMA and DMD. This novel device can serve as a more affordable and versatile measurement instrument for neuromuscular disorders that affect gait and balance. All participants will be observed and measured while wearing the instrumented insoles in the lab and in real-life environments.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following categories:

   * Genetic confirmation of spinal muscular atrophy
   * Genetic confirmation of Duchenne or Becker muscular dystrophy or evidence on muscle biopsy with a clinical presentation consistent with DMD/BMD
   * Healthy individuals.
2. Able to walk independently at least 25 meters

Exclusion Criteria:

1. Unable to walk 25 meters independently.
2. Use of investigational medications intended for the treatment of SMA or DMD/BMD within 30 days prior to study entry.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study sample will include 13 ambulatory SMA participants, 13 ambulatory DMD participants, and 13 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Validation of Instrumented Insoles: Six Minute Walk Test | Baseline
  To measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway participants will complete the Six Minute Walk Test. This test is an objective evaluation of functional exercise capacity, measures the maximum distance a person can walk in six minutes over a 25 meter course. This will be performed in a corridor and include the instrumented walkway.
Validation of Instrumented Insoles: 10 Meter Walk/Run | Baseline
  To measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway, participants will walk, or run if able to, for 10 meters on the instrumented walkway.
Validation of Instrumented Insoles: Time Up and Go Test (TUG) | Baseline
  To measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway, participants will complete the TUG test. This test is designed to test mobility after a person stands up from a seated position. This will be completed on the instrumented walkway.
Validation of Instrumented Insoles: Straight Line Walking | Baseline
  To measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway, participants will be asked to walk in a straight line multiple times over the instrumented walkway.
Validation of Instrumented Insoles: Circle Walking | Baseline
  To measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway participants will be asked to walk a series of half-circles on the instrumented walkway.
Muscle Strength Testing with Hand-held Dynamometry (HHD) | Baseline
  HHD is used to assess strength of selected muscles.

SECONDARY OUTCOMES:
Free-living Testing of Instrumented Insoles | One week
  To determine spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity using instrumented insoles, 5 participants with SMA, 5 participants with DMD, and 5 healthy controls will be asked to wear the insoles along with a validated activity tracker. Participants will be asked to wear the insoles during a visit to the lab, and then for one week at home in a real-life environment. Participants will be asked to wear the insoles and activity tracker for at least 4 hours per day when at home.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Montes, PT, EdD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Montes J, Kanner CH, Duong T, Rodriguez-Torres R, Uher D, Young SD, Farooquee R, Druffner A, Pasternak A, Fragala-Pinkham M, Zanotto D. Wearable-Derived Patterns of Performance Fatigability During Gait in Spinal Muscular Atrophy. Muscle Nerve. 2025 Sep;72(3):493-501. doi: 10.1002/mus.28461. Epub 2025 Jun 25. PMID 40557477